

## Tour de Borobudur Troponin Study on Predictors and Synergistic Role of MDA and Hs-CRP Levels (TdBTS)

## Tour de Borobudur Troponin Study

ClinicalTrials.gov Identifier: NCT03310450

## **Statistical Analysis**

12th October 2017

Tour de Borobudur Troponin Study on Predictors and Synergistic Role of MDA and Hs-CRP Levels (TdBTS)

Tour de Borobudur Troponin Study

ClinicalTrials.gov Identifier: NCT03310450

**Statistical Analysis** 

All data were reported as mean ± standard deviation (SD) [range] unless stated otherwise, and

statistical significance was assumed at a p-value < 0.05. Statistical analyses were performed using the

Statistical Package for the Social Sciences (IBM SPSS Statistics for Windows, Version 23.0, IBM Corp.,

NY, USA). The normality of the data distribution was examined by the Kolmogorov–Smirnov test. When

the data demonstrated a non-Gaussian distribution, natural logarithmic transformation was applied. Paired

Student's t-test was used to test the significance of the differences between the group with cTnI elevation

and post-touring levels for continuously distributed data. A backward stepwise binary logistic regression

analysis was used to identify factors that were significantly related to post-exercise cTnI elevation. Based

on our hypothesis, we included age, BMI, medical history, total and HDL cholesterol, leucocyte indices,

and HR in our model as potential determinants to predict post-exercise cTnI level. Thereafter, all predictors

with a p-value < 0.25 were retained in the final regression model. Binary logistic analysis was used to

determine the predictor most related to cTnI elevation.